CLINICAL TRIAL: NCT02224794
Title: LIFE Study: Least Invasive Fast-Track EVAR With the Ovation® Abdominal Stent Graft Platform
Brief Title: LIFE Study: Least Invasive Fast-Track EVAR
Status: Completed | Type: Observational
Sponsor: TriVascular, Inc. (Industry)
Responsible Party: Sponsor
Organization: Endologix (Industry)
Other Study IDs: 771-0014
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal; aortic; aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Fast-Track Group: includes subjects who complete the Fast-Track EVAR protocol
  Interventions: Device: Ovation® Abdominal Stent Graft Platform
- Standard P-EVAR Group: includes subjects who do not complete the Fast-Track EVAR protocol, and their procedures are completed with bilateral percutaneous access
  Interventions: Device: Ovation® Abdominal Stent Graft Platform
- Standard EVAR Group: includes subjects who do not complete the Fast-Track EVAR protocol, and their procedures are not completed with bilateral percutaneous access (i.e. converted to femoral cutdown or open surgical repair)
  Interventions: Device: Ovation® Abdominal Stent Graft Platform

INTERVENTIONS:
Device: Ovation® Abdominal Stent Graft Platform

SUMMARY:
The primary objectives of the LIFE Study are to demonstrate the clinical and cost benefits associated with using the Ovation® Abdominal Stent Graft Platform under the least invasive conditions defined in the Fast-Track EVAR protocol. The key elements of the Fast-Track EVAR protocol include: appropriate patient selection, bilateral percutaneous access, no general anesthesia, no ICU admission post procedure, and next day discharge.

DETAILED DESCRIPTION:
The LIFE Study is a prospective, consecutively enrolling, non-randomized multi center post-market registry to evaluate the ultra low profile (14F) Ovation Abdominal Stent Graft Platform when using in the Percutaneous Endovascular Aneurysm Repair (P-EVAR) treatment of patients with AAA using a Fast-Track EVAR protocol.

250 study patients will be enrolled at up to 40 institutions. Follow-up period is one month.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age.
* Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study).
* Patient has signed an IRB approved informed consent form.
* Patient is considered by the treating physician to be a candidate for elective open surgical repair of the AAA.
* Patient has an infrarenal abdominal aortic aneurysm that meets at least one of the following: abdominal aortic aneurysm >5.0 cm in diameter, aneurysm has increased in size by 0.5 cm in last 6 months, or maximum diameter of aneurysm exceeds 1.5 times the transverse dimension of an adjacent non-aneurysm exceeds 1.5 times the transverse dimension of an adjacent non-aneurysmal aortic segment.
* Patient has suitable anatomy that allows use of the TriVascular Ovation® Abdominal Stent Graft Platform.
* Patient has suitable femoral arteries at the percutaneous access site that allow use of the Perclose ProGlide Suture-Mediated Closure System via the pre-close technique.
* Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria:

* Patient has a need for emergent surgery.
* Patient has a dissecting aneurysm.
* Patient has an acutely ruptured aneurysm.
* Patient has an acute vascular injury.
* Patient has had a previous repair of the abdominal aortic aneurysm or the iliac artery.
* Patient has a mycotic aneurysm or has an active systemic infection.
* Patient has unstable angina.
* Patient has unstable peripheral artery disease with critical limb ischemia.
* Patient has congestive heart failure.
* Patient has had a myocardial infarction and/or stroke within the past 3 months.
* Patient requires use of techniques that would cover the renal arteries.
* Patient requires planned adjunctive devices to complete the procedure.
* Patient has a major surgical or interventional procedure planned during or within ±30 days of the AAA repair.
* Patient has history of connective tissue disease.
* Patient has history of bleeding disorders or refuses blood transfusions.
* Patient has dialysis dependent renal failure or baseline serum creatinine level >2.0mg/dl.
* Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
* Patient has a known allergy or intolerance to polytetrafluoroethylene (PTFE), PEG-based polymers, fluorinated ethylene propylene (FEP) or nitinol.
* Patient is on home oxygen.
* Patient is morbidly obese (BMI ≥40 kg/m2).
* Patient was admitted from a skilled nursing facility.
* Patient has a limited life expectancy of less than 1 year.
* Patient has an inability to be discharged within 1 day of the procedure.
* Patient is currently participating in an investigational device or drug clinical trial.
* Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll male and female subjects 18 years and older that have an AAA and meet all other inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Major Adverse Events | 30 days

SECONDARY OUTCOMES:
Serious and non-serious adverse events, including vascular and major access site vascular complications | 30 days
Assess technical success, defined as percent of procedures successfully completed with bilateral percutaneous access | 30 days
Treatment success, defined as percent of subjects who successfully follow least invasive protocol through discharge | 30 days
Blood loss, including if transfusion required | 30 days
Percent of procedures completed without general anesthesia | 30 days
Anesthesia time | 30 days
Procedure time | 30 days
Contrast volume | 30 days
Fluoroscopy time | 30 days
Time to hemostasis | 30 days
Time to ambulation | 30 days
Time to normal diet | 30 days
Groin pain | 30 days
Quality of Life | 30 days
Percent of subjects discharged without ICU admission | 30 days
Length of ICU stay, if required | 30 days
Length of hospital stay | 30 days
Percent of subjects discharged within only one midnight stay | 30 days
Freedom from type I and III endoleaks | 30 days
Freedom from AAA rupture | 30 days
Freedom from conversion to open repair | 30 days
Freedom from AAA related secondary interventions | 30 days
Freedom from mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Zvonimir Krajcer, MD, Principal Investigator — CHI St. Luke's Health, Texas; Venkatesh Ramaiah, MD, Principal Investigator — Arizona Heart Institute
Locations (2):
- United States (2):
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - St. Luke's Episcopal Hospital, Houston, Texas

REFERENCES:
- [Derived] Krajcer Z, Ramaiah VG, Henao EA, Metzger DC, Nelson WK, Moursi MM, Rajasinghe HA, Al-Dallow R, Miller LE; LIFE Registry Investigators. Perioperative Outcomes From the Prospective Multicenter Least Invasive Fast-Track EVAR (LIFE) Registry. J Endovasc Ther. 2018 Feb;25(1):6-13. doi: 10.1177/1526602817747871. Epub 2017 Dec 18. PMID 29251207
- [Derived] Krajcer Z, Ramaiah V, Huetter M. Fast-track endovascular aneurysm repair: rationale and design of the multicenter Least Invasive Fast-Track EVAR (LIFE) registry. BMC Cardiovasc Disord. 2015 Dec 19;15:174. doi: 10.1186/s12872-015-0167-1. PMID 26685936
- See also: Related Info — http://www.endologix.com